CLINICAL TRIAL: NCT00103298
Title: A Phase II Trial of Isolated Hepatic Perfusion (IHP) and Systemic FOLFOX4 for Subjects With Metastatic Unresectable Colorectal Cancers of the Liver With ≥ 40% Hepatic Tumor Burden
Brief Title: Isolated Hepatic Perfusion With Melphalan Followed by Combination Chemotherapy in Treating Patients With Unresectable Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000409754; NCI-05-C-0025; NCT00096889 (obsolete NCT alias)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2006-02

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Melphalan; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: isolated perfusion
Drug: leucovorin calcium
Drug: melphalan
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, leucovorin, oxaliplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving the drugs in different ways may kill more tumor cells.

PURPOSE: This phase II trial is studying how well isolated hepatic perfusion with melphalan followed by combination chemotherapy works in treating patients with unresectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response and duration of response in patients with previously untreated unresectable liver metastases secondary to colorectal cancer treated with isolated hepatic perfusion with melphalan followed by leucovorin calcium, oxaliplatin, and fluorouracil.

Secondary

* Determine the patterns of recurrence (liver vs systemic) in patients treated with this regimen.
* Determine progression-free and overall survival of patients treated with this regimen.
* Correlate health-related quality of life with length of survival of patients treated with this regimen.

OUTLINE: Patients undergo exploratory laparotomy. Patients with evidence of carcinomatosis not previously visualized on scans but found on surgical exploration are removed from the study. All other patients then undergo isolated hepatic perfusion (IHP). Once IHP is established, melphalan is administered intra-arterially over 3-5 minutes and then circulated throughout the liver for 1 hour. Approximately 6-12 weeks later, patients receive systemic chemotherapy comprising oxaliplatin IV over 2 hours on day 1 and leucovorin calcium IV over 2 hours and fluorouracil IV continuously over 22 hours on days 1-2. Courses with systemic chemotherapy repeat every 14 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, after laparotomy, after completion of systemic chemotherapy, and then every 6 months thereafter.

After completion of study treatment, patients are followed every 3 months for 1 year, every 3-4 months for 2 years, and then every 6 months until disease progression.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal cancer

  * Metastatic disease limited to the parenchyma of the liver

    * No evidence of unresectable extrahepatic disease by preoperative radiology

      * Limited extra-hepatic disease and dominant life-limiting liver disease allowed provided extra-hepatic sites are treatable by local ablative measures (e.g., surgical resection or external beam radiotherapy)
* At least 40% hepatic replacement by tumor by axial CT scan or MRI
* Unresectable liver metastases, defined by 1 of the following:

  * More than 3 sites of disease in the liver
  * Bilobar disease
  * Tumor abutting major vascular or ductal structures
* Measurable disease
* Previously untreated disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Hematocrit > 27.0%
* WBC > 3,000/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 2.0 mg/dL
* PT < 2 seconds above upper limit of normal
* Elevated transaminase levels allowed if due to liver metastases
* No cirrhosis by biopsy
* No significant portal hypertension as manifested by any of the following:

  * Ascites
  * Esophageal varices by endoscopy
  * Significant collateral vessels around the organs drained by the portal venous system by radiography
* No chronic active hepatitis

  * Hepatitis B and C surface antigen negative
* No history of veno-occlusive disease

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No ischemic cardiac disease
* No history of congestive heart failure
* LVEF > 40% by echocardiogram or stress thallium scan (for patients with cardiac disease)

Pulmonary

* No chronic obstructive pulmonary disease or other chronic pulmonary disease
* Pulmonary function tests ≥ 50% of predicted (for patients with pulmonary disease)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight > 30 kg
* No active infection
* No peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior adjuvant chemotherapy (including leucovorin calcium, oxaliplatin, and fluorouracil) allowed provided it was administered > 6 months before liver metastases were diagnosed

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy for this malignancy and recovered

Surgery

* Not specified

Other

* No concurrent chronic anticoagulation therapy
* No concurrent immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Response and duration of response

SECONDARY OUTCOMES:
Patterns of recurrence
Progression-free and overall survival
Correlation of health-related quality of life with length of survival

CONTACTS AND LOCATIONS:
Overall Officials: H. Richard Alexander, MD, FACS, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States